CLINICAL TRIAL: NCT05316168
Title: Isolated Adductor Canal Block vs Adductor Canal Block With IPACK in ACL Reconstruction: A Randomized, Prospective Trial
Brief Title: Post Operative Pain Management for ACL Reconstruction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ftjo21D.1099
Record Dates: First submitted 2021-12-02; First posted 2022-04-07 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Dexamethasone; oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- isolated adductor canal block (ACB) (Active Comparator): Adductor Canal Block with 20cc 0.5% bupivacaine HCl + 2mg dexamethasone.
  Interventions: Drug: Bupivacaine HCl 0.5% Injectable Solution; Drug: Dexamethasone; Drug: Percocet 5Mg-325Mg Tablet
- isolated adductor canal block (ACB) + IPACK (Active Comparator): ACB with 20cc 0.5% bupivacaine HCl + 2mg dexamethasone, and iPACK with 20cc 0.5% bupivacaine + 2mg dexamethasone.
  Interventions: Drug: Bupivacaine HCl 0.5% Injectable Solution; Drug: Dexamethasone; Procedure: Infiltration between Popliteal Artery and Capsule of the knee (iPACK); Drug: Percocet 5Mg-325Mg Tablet

INTERVENTIONS:
Drug: Bupivacaine HCl 0.5% Injectable Solution — During adductor canal block participants will receive 20cc of Bupivacaine HCl 0.5%
Drug: Dexamethasone — During adductor canal block participants will receive 2mg Dexamethasone
Procedure: Infiltration between Popliteal Artery and Capsule of the knee (iPACK) — Prior to closing the surgical wound participants will receive a local injections of 20cc 0.5% bupivacaine mixed with 2mg dexamethasone
  Arms: isolated adductor canal block (ACB) + IPACK
Drug: Percocet 5Mg-325Mg Tablet — Participant will receive 20 Percocet 5/325mg tablets post surgery for pain control

SUMMARY:
Health care providers are seeking methods to limit post-operative pain and opioid prescriptions to reduce the burden of the national opioid use epidemic. Adductor canal block (ACB) is a peripheral nerve block that has been shown to reduce pain and opioid usage with minimal effect on quadriceps function in patients undergoing arthroscopic knee surgery. Infiltration between Popliteal Artery and Capsule of the Knee (iPACK) block has also shown promise in reducing pain and opioid usage, specifically reducing posterior knee pain, which ACB is not able to achieve. To our knowledge, there is currently no study in the orthopedic literature comparing post-operative pain and opioid consumption in ACL reconstruction (ACLR) patients who received isolated ACB versus ACB with IPACK.

The primary aim of this study is to investigate the role of IPACK in combination with ACB in reducing peri-operative (14-days) pain levels in ACLR patients. The secondary aim is to determine the effectiveness of IPACK in reducing post-operative opioid use. The tertiary aim is to determine any effect of IPACK on post-operative functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing primary ACLR for ACL tear, including patients with concomitant meniscectomy or meniscal repair.

Exclusion Criteria:

* Revision ACLR, worker's compensation, pregnancy, age<18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Post operative pain management | 14 days
  This will be measured by the participants completing a pain and medication Use questionnaire
Post operative pain management 2 | 6 months
  Participants will also complete the International Knee Documentation Committee (IKDC) questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States